CLINICAL TRIAL: NCT05423275
Title: Light and Ion Maintenance In Treatment for Depression (LIMIT-D): Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Toronto (Other); Université de Montréal (Other); Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other); Ontario Brain Institute (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Raymond Lam, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H22-01067
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder, Recurrent, in Remission
Keywords: antidepressants; discontinuation; relapse prevention; light therapy; negative ions; depression
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depression | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Randomized, two-group, parallel, relapse prevention design
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and the clinical outcome assessor is masked as to whether the study device is active or inactive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative ion therapy (Active Comparator): High density negative ions at 3.4 trillion ions per second with no detectable ozone, used for 30 minutes as soon as possible after awakening, preferably between 7:00-8:00 am.
  Interventions: Device: Negative ion therapy
- Light therapy (Active Comparator): 4000 Kelvin white fluorescent light rated at 10,000 lux at 14 inches from screen to cornea, with an ultraviolet filter, used for 30 minutes as soon as possible after awakening, preferably between 7:00-8:00 am.
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Negative ion therapy — Negative ion generator
  Arms: Negative ion therapy
Device: Light therapy — Fluorescent light box
  Arms: Light therapy

SUMMARY:
Antidepressants are widely used as first-line treatments for major depressive disorder (MDD). Clinical guidelines recommend 6-24 months of "maintenance" antidepressant treatment, after patients achieve symptom remission, to prevent relapse but many people stop antidepressants too soon relapse into another depressive episode. We will test non-medication treatments, negative ion therapy and light therapy, to see they can substitute for antidepressants to prevent relapse. This is a "feasibility" study to see if participants use study treatments properly, before doing a larger, definitive trial. In this 28-week study, 100 participants with MDD who are in remission with antidepressants will be treated with light therapy or negative ion therapy (with half of devices active and half inactive) while slowly discontinuing the antidepressant, and monitored for relapse.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of a multicentre, randomized, trial of light therapy and negative ion therapy as substitutes for antidepressants for maintenance treatment for patients with recurrent major depressive disorder (MDD).

The study design for this feasibility study mirrors the full LIMIT-D protocol: a 28-week, double-blind (participant and outcome rater) relapse prevention study with 100 participants randomized 1:1 to one of two study treatments, light therapy or negative ion therapy, and assessed for relapse over 28 weeks. Half the study devices are modified to be inactive. After 2 weeks of study treatment, the participant's antidepressant will be tapered and discontinued between Week 2 and Week 8.

Participants are assessed for relapse at each scheduled study visit (every 2 weeks during antidepressant taper until week 8, then every 4 weeks until end of study treatment at Week 28) by blind outcome raters. In addition, they complete an online Personal Health Questionnaire (PHQ-9) self-rated depression symptom scale bi-weekly; if total score is 10 or higher OR the suicide item score is 2 or higher, participants are booked for a relapse-assessment visit and relapse-verification study visit at least 1 week apart. Relapse will be defined as any of the following:

1. MADRS total score 20 or higher for at least 2 consecutive weeks and Diagnostic and Statistical Manual (DSM-5) criteria for major depressive episode at the Relapse-Verification visit.
2. Hospitalization for worsening of depression.
3. Suicidal ideation with intent or plan, or suicidal behaviour.
4. Any change in treatment for depression (e.g., starting an antidepressant).

At each visit, clinician-rated and self-rated symptom, side effect, and functioning measures are completed. The primary feasibility outcome is recruitment rate; secondary feasibility outcomes include adherence to study treatment, successful discontinuation of antidepressants rate, and all-cause dropout rate. Secondary clinical outcomes include relapse rate, time to relapse, adverse events, and safety profiles.

Participants will wear an actigraph at home during the 28-week study treatment period to assess sleep, light and activity/circadian rhythms. There is a final observational visit by Zoom videoconference at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM-5) criteria for MDD, as determined by the Structured Clinical Interview for DSM-5 (SCID).
* Taking a first-line antidepressant at approved doses (Table 1), with dose unchanged in the past month.
* Participant desire to discontinue antidepressant treatment because of adverse effects or other reasons;
* In remission as defined by score ≤10 on the clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) at both the screening visit and baseline visit, at least 2 weeks apart.
* Willing and able to complete self-report and online assessments including sufficient fluency in English or French.

Exclusion Criteria:

* Any psychiatric diagnosis other than MDD that is considered the primary diagnosis, including Bipolar I or Bipolar-II (lifetime). Note that comorbid anxiety disorders (e.g., generalized anxiety disorder, social anxiety disorder) will not be excluded if the anxiety disorder is not the primary diagnosis.
* Diagnosis of MDD with seasonal pattern (i.e., seasonal affective disorder, SAD) or with psychotic features (lifetime).
* Significant personality disorder diagnosis [e.g., antisocial] by MINI and clinical assessment.
* High suicidal risk, defined by clinician judgment.
* History of alcohol or substance use disorder, with a severity of at least moderate or severe, within 6 months before screening.
* Significant neurological disorders, head trauma, or other unstable medical conditions.
* Regular use of psychotropic medication other than an antidepressant or benzodiazepines (e.g., antipsychotics, mood stabilizers); Note - Stimulant medications for Attention-Deficit Hyperactivity Disorder are allowed if dose is stable in past month.
* History of severe antidepressant discontinuation effects.
* Retinal disease or other eye condition (e.g., macular degeneration) precluding the use of bright light treatment.
* Use of photosensitizing medication (thioridazine, chloroquine, 8-methoxypsoralen) within 1 week of baseline visit.
* Initiated formal psychotherapy (e.g., cognitive-behavioural therapy) within 3 months of Visit 1, or who plan to initiate psychotherapy during the study.
* Continued use of any other evidence-based treatment for depression.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 36 months
  The number of participants entered into the study during the recruitment period.

SECONDARY OUTCOMES:
Adherence to study treatment | 28 weeks
  Percentage of scheduled time that participants use the study treatment
Rate of stopping antidepressants | 8 weeks
  Rate of success in tapering and discontinuing antidepressants
All-cause dropout rate | 28 weeks
  Rate of dropouts from the study for any cause

OTHER OUTCOMES:
Time to relapse | 28 weeks
  Time to protocol-defined relapse, based on survival analysis
Relapse rate | 28 weeks
  Rate of relapses, based on survival analysis
Adverse events | 28 weeks
  Number and severity of adverse events
Serious adverse events | 28 weeks
  Number of serious adverse events including hypomanic mood switch

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W Lam, MD, Principal Investigator — University of British Columbia
Locations (1):
- Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia, Canada